CLINICAL TRIAL: NCT05643573
Title: A Multicenter, International, Randomized, Active Comparator-controlled, Double-blind, Double-dummy, Parallel-group, 2-arm, Phase 3 Study to Compare the Efficacy and Safety of the Oral FXIa Inhibitor Asundexian (BAY 2433334) With Apixaban for the Prevention of Stroke or Systemic Embolism in Male and Female Participants Aged 18 Years and Older With Atrial Fibrillation at Risk for Stroke
Brief Title: A Study to Learn How Well the Study Treatment Asundexian Works and How Safe it is Compared to Apixaban to Prevent Stroke or Systemic Embolism in People With Irregular and Often Rapid Heartbeat (Atrial Fibrillation), and at Risk for Stroke
Acronym: OCEANIC-AF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Independent Data Monitoring Committee (IDMC) recommendation to stop the study
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19767; 2023-503794-38-00 (Other: CTIS (EU)); 2022-000758-28 (EudraCT Number)
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Prevention of Stroke or Systemic Embolism; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — asundexian; apixaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Asundexian (Experimental): Participants will receive asundexian and apixaban matching placebo.
  Interventions: Drug: Asundexian (BAY2433334); Drug: Apixaban matching placebo
- Apixaban (Active Comparator): Participants will receive apixaban and asundexian matching placebo.
  Interventions: Drug: Apixaban; Drug: Asundexian matching placebo

INTERVENTIONS:
Drug: Asundexian (BAY2433334) — Once a day
  Arms: Asundexian
Drug: Apixaban — 5 mg or 2.5 mg, twice a day, according to product label.
  Arms: Apixaban
Drug: Asundexian matching placebo — Placebo to asundexian, once a day
  Arms: Apixaban
Drug: Apixaban matching placebo — Placebo to apixaban, twice a day
  Arms: Asundexian

SUMMARY:
Researchers are looking for a better way to treat people with atrial fibrillation (AF) and prevent stroke or systemic embolism (blood clots travelling through the blood stream to plug another vessel).

Atrial fibrillation is a condition of having irregular and often rapid heartbeat. It can lead to the formation of blood clots in the heart which can travel through the blood stream to plug another vessel, and like this lead to serious and life-threatening conditions, such as a stroke. A stroke occurs because the brain tissue beyond the blockage no longer receives nutrients and oxygen so that brain cells die. As strokes arising from atrial fibrillation can involve extensive areas of the brain, it is important to prevent them.

Blood clots are formed in a process known as coagulation. Medications are already available to prevent the formation of blood clots. When taken by mouth (orally), they are known as oral anticoagulants (OACs) including apixaban. OACs decrease the risk of the above-mentioned serious and life-threatening conditions. The main side effect of OACs is an increase of the risk of bleeding.

The study treatment asundexian is a new type of anticoagulant currently under development to provide further treatment options. Asundexian aims to further improve the standard of care with regard to the risk of bleeding.

The main purpose of this study is to collect more data about how well asundexian works to prevent stroke and systemic embolism and how safe it is compared to apixaban in people with atrial fibrillation and at high risk for stroke.

To see how well the study treatment asundexian works researchers compare:

* how long asundexian works well and
* how long apixaban works well after the start of the treatment. Working well means that the treatments can prevent the following from happening:
* stroke and/or
* systemic embolism. The study will keep collecting data until a certain number of strokes or embolisms happen in the study.

To see how safe asundexian is, the researchers will compare how often major bleedings occur after taking the study treatments asundexian and apixaban, respectively. Major bleedings are bleedings that have a serious or even life-threatening impact on a person's health.

The study participants will be randomly (by chance) assigned to 1 of 2 treatment groups, A and B. Dependent on the treatment group, the participants will either take the study treatment asundexian by mouth once a day or apixaban by mouth twice a day for approximately 9 - 33 months.

Each participant will be in the study for approximately 9 - 34 months. There will be visits to the study site every 3 to 6 months and up to 7 phone calls. Those participants who do not want or are unable to have visits to the study site may join the study remotely in selected locations. The location name contains the abbreviation - DCT in such cases.

During the study, the study team will:

* take blood samples
* do physical examinations
* examine heart health using an electrocardiogram (ECG)
* check vital signs such as blood pressure and heart rate
* do pregnancy tests
* ask the participants questions about their quality of life
* ask the participants questions about how they are feeling and what adverse events they are having.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* The patient willing and able to understand the Patient information Sheet and provide written informed consent
* Atrial fibrillation with an indication for indefinite treatment with an oral anticoagulant
* CHA2DS2-VASc score ≥ 3 if male or ≥ 4 if female, OR CHA2DS2-VASc score of 2 if male or 3 if female and at least one of the following enrichment criteria:

  * age ≥ 70
  * previous stroke, transient ischemic attack, or systemic embolism
  * renal dysfunction with eGFR < 50 ml/min within 14 days prior to randomization
  * prior episode of non-traumatic major bleeding
  * current single agent antiplatelet therapy planned to continue for at least 6 months after randomization
  * ≤ 6 consecutive weeks of treatment with oral anticoagulant prior to randomization.

Exclusion Criteria:

* Mechanical heart valve prosthesis
* Moderate-to-severe mitral stenosis at the time of study inclusion.
* Atrial fibrillation only due to reversible cause.
* Participants after successful ablation therapy without documented recurrent AF or participants after left atrial appendage occlusion / exclusion or plan for ablation or Left atrial appendage (LAA) occlusion / exclusion within the next 6 months.
* Recent ischemic stroke (within 7 days prior to randomization).
* Active non-trivial bleeding; known chronic bleeding disorder ; history of non-traumatic intracranial hemorrhage.
* Known significant liver disease or known hepatic insufficiency classified as Child-Pugh B or C at randomization.
* Estimated glomerular filtration rate (eGFR) < 25 mL/min/1.73 m2 within 14 days prior to randomization or on dialysis or expected to be started on dialysis within the next 12 months starting from randomization.
* Major surgery during the last 30 days prior to randomization.
* Known allergy, intolerance or hypersensitivity to either of the study interventions.
* Any contraindication for the use of an anticoagulant or listed in the local labelling for apixaban.
* Requirement for chronic anticoagulation for a different indication than AF, e.g. mechanical heart valve or left ventricular cardiac thrombus (atrial thrombus is allowed), or dual antiplatelet therapy (single agent therapy is allowed).
* Treatment with Vitamin K antagonist (VKA) in the 10 days prior to randomization.
* Concomitant use of or anticipated need for:

  * daily or near daily (> 5 days per week) therapy with nonsteroidal anti-inflammatory drugs (NSAIDs) for more than 4 weeks during the study
  * herbal or traditional medicine, and / or supplements with known anticoagulant and / or antiplatelet effect
  * combined P-glycoprotein (P-gp) and strong cytochrome P450 isoenzyme 3A4 (CYP3A4) inhibitors
  * combined P-gp and strong / moderate CYP3A4 inducers Respective substances (apart from NSAIDs) must be stopped - in case of combined inhibitors / inducers of CYP3A4 and P-gp for at least 14 days before randomization.
* Previous (within 30 days or 5 half-lives of the investigational drug, whichever is longer) or concomitant participation in another clinical study with investigational medicinal product(s) or device(s). Registries and observational studies are allowed.
* Known current alcohol and / or illicit drug abuse.
* Close affiliation with the investigational site.
* Any other history, condition or therapy, or uncontrolled intercurrent illness which would make the participant unsuitable for the study vulnerable or life expectancy < 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14830 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1069):
- United States (163):
  - SEC Clinical Research, Dothan, Alabama
  - Eastern Shore Research Institute, LLC | Fairhope, AL, Fairhope, Alabama
  - Mobile Heart Specialists, PC, Mobile, Alabama
  - University of South Alabama Medical Center, Mobile, Alabama
  - Arkansas Cardiology | Little Rock, Little Rock, Arkansas
  - Valley Clinical Trials, Inc. | Covina, CA, Covina, California
  - Science 37, Culver City, California
  - University of California, Irvine, Irvine, California
  - VA Long Beach Healthcare System, Long Beach, California
  - VA Greater Los Angeles Healthcare System | West Los Angeles VA Medical Center - Cardiology Department, Los Angeles, California
  - Radin Cardiovascular Medical Group, Newport Beach, California
  - Amicis Research Center | Northridge, CA, Northridge, California
  - Cottage Health | Santa Barbara Cottage Hospital - Cardiology Department, Santa Barbara, California
  - NorthBay Clinical Research, LLC | Santa Rosa, CA, Santa Rosa, California
  - The Lundquist Institute | Cardiology Department, Torrance, California
  - Harbor - UCLA Medical Center, Torrance, California
  - Blue Coast Research Center, LLC, Vista, California
  - Interventional Cardiology Medical Group | West Hills, CA, West Hills, California
  - University of Colorado Hospital - Cardiology, Aurora, Colorado
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Cardiology Associates of Fairfield County, P.C. | Stamford, CT, Norwalk, Connecticut
  - Integrity Clinical Research | Florida Premier Cardiology, Boynton Beach, Florida
  - Integrity Clinical Research | Cardiology Associates of South Florida, Boynton Beach, Florida
  - Cardiovascular & Vein Center of Florida | Bradenton, FL, Bradenton, Florida
  - Nova Clinical Research | Brandenton, FL, Bradenton, Florida
  - Clearwater Cardiovascular Associates | Clearwater, FL, Clearwater, Florida
  - Cardiology Consultants, PA, Daytona Beach, Florida
  - Cardiology Associates Research Company, Daytona Beach, Florida
  - Integrity Clinical Research | Heller Heart Health, Delray Beach, Florida
  - North Florida Foundation For Research And Education | Veterans Benefits Administration, Gainesville, Florida
  - Indago Research and Health Center | Hialeah, FL, Hialeah, Florida
  - Encore Research Group | Nature Coast Clinical Research - Inverness, Inverness, Florida
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Heart Vein & Vascular | Longwood, FL, Longwood, Florida
  - Life Spring Research | Miami, FL, Miami, Florida
  - Southwest Florida Research | Naples, FL, Naples, Florida
  - Advanced Research for Health Improvement, LLC | Naples, FL, Naples, Florida
  - Cardiology Partners Clinical Research Institute | Palm Beach Gardens Office, Palm Beach Gardens, Florida
  - Baptist Heart and Vascular/Cardiology Consultants, Pensacola, Florida
  - Peace River Cardiovascular Center | Port Charlotte, FL, Port Charlotte, Florida
  - Encore Research Group | St. Johns Center for Clinical Research, Saint Augustine, Florida
  - East Coast Institute for Research | St. Augustine, FL, Saint Augustine, Florida
  - Cardiovascular Center of Sarasota Foundation for Research and Education | Sarasota, FL, Sarasota, Florida
  - Cardiology Partners Clinical Research Institute | Wellington Office, Wellington, Florida
  - St. Mary's Medical Center | West Palm Beach - Neurology Department, West Palm Beach, Florida
  - Morehouse School of Medicine | Clinical Research Centre, Atlanta, Georgia
  - NSC Cardiology | Johns Creek, GA, Cumming, Georgia
  - Alta Pharmaceutical Research Center, LLC, Peachtree Corners, Georgia
  - Atlanta Heart Specialists, LLC, Tucker, Georgia
  - St. Luke's Health System | St. Luke's Clinic - Idaho Cardiology Associates, Meridian, Idaho
  - Northwestern University, Chicago, Illinois
  - Northshore Medical Center, Glenview, Illinois
  - Affinity Health Research Institute | Oak Brook, IL, Oak Brook, Illinois
  - Midwest Cardiovascular Research and Education Foundation | Elkhart, IN, Elkhart, Indiana
  - Cardiovascular Research of Northwest Indiana, LLC. | Munster, IN, Hammond, Indiana
  - IU Health Physicians Cardiology, Indianapolis, Indiana
  - Reid Physician Associates | Cardiology Department, Richmond, Indiana
  - Accellacare | Ames, IA, Ames, Iowa
  - University of Iowa, Iowa City, Iowa
  - Kansas Nephrology Physicians, PA, Wichita, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Medical Group - Louisville Cardiology, Louisville, Kentucky
  - Research Integrity, LLC, Owensboro, Kentucky
  - Cambridge Medical Trials, Alexandria, Louisiana
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - Cardiovascular Associates Research, LLC, Covington, Louisiana
  - Ochsner Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana Heart Center Research - Slidell, Slidell, Louisiana
  - Northeast Cardiology Associates, Bangor, Maine
  - MaineHealth Maine Medical Center | Maine Medical Partners Cardiology, Scarborough, Maine
  - LifeBridge Health | Sinai Hospital - Platelet and Thrombosis Research Department, Baltimore, Maryland
  - Spectrum Clinical Research | Maryland Cardiovascular Specialists, Baltimore, Maryland
  - Johns Hopkins Hospital/Health System, Baltimore, Maryland
  - Johns Hopkins University School of Medicine | CAPRES, Columbia, Maryland
  - Anderson Medical Group and Cardiology | Anderson Medical Research, LLC, Ft. Washington, Maryland
  - Adventist HealthCare | White Oak Medical Center, Silver Spring, Maryland
  - McLaren Health Care | McLaren Bay Region - Research Department, Bay City, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - AA Medical Research Center | Flint, MI, Flint, Michigan
  - Sparrow Clinical Research Institute | Sparrow Hospital - Clinical Research Department, Lansing, Michigan
  - M Health Fairview, Maplewood, Minnesota
  - Veterans Benefits Administration | Minneapolis VA Medical Center - Cardiology Department, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Minneapolis Heart Institute, Saint Paul, Minnesota
  - Jackson Heart Clinic | Jackson, MS, Jackson, Mississippi
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - St. Louis Heart & Vascular, PC, St Louis, Missouri
  - CHI Health Clinic Heart Institute - Grand Island, Grand Island, Nebraska
  - Advanced Heart Care, LLC | Bridgewater, NJ, Bridgewater, New Jersey
  - NJ Heart | Linden, NJ, Linden, New Jersey
  - Garden State Heart Care, Manalapan, New Jersey
  - Inspira Medical Centers | Clinical Research Office, Mullica Hill, New Jersey
  - The Valley Hospital, Inc., Ridgewood, New Jersey
  - Cooper Specialty Care at Voorhees, Voorhees Township, New Jersey
  - IMA Clinical Research | Warren, NJ, Warren Township, New Jersey
  - Circuit Clinical/Crystal Run, Middletown, New York
  - NYU Langone Health | NYU Langone Medical Associates Chelsea - Cardiovascular Research, New York, New York
  - Division of Cardiovascular Research at Peconic Bay Med Ctr, Riverhead, New York
  - Great Lakes Medical Research | Westfield, NY, Westfield, New York
  - University of North Carolina at Chapel Hill | Cardiology Department, Chapel Hill, North Carolina
  - Duke University | Duke Clinical Research Institute - Participant Research Operations, Durham, North Carolina
  - Duke Univ. Medical Center, Durham, North Carolina
  - Medication Management | Greensboro - Cardiology, Greensboro, North Carolina
  - Clinical Trials of America, Inc., Mount Airy, North Carolina
  - Lillestol Research LLC | Fargo, ND, Fargo, North Dakota
  - Aultman | Aultman Hospital Main Campus - Clinical Trials, Canton, Ohio
  - Kettering Health Network | Research Institute, Kettering, Ohio
  - Rama Research LLC | Marion, OH, Marion, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - South Oklahoma Heart Research, LLC, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Capital Area Research | Camp Hill, PA, Camp Hill, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - University of Pittsburgh Medical Center, Hamot | Clinical Trials and Research, Erie, Pennsylvania
  - Pennsylvania State University College of Medicine, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Einstein Healthcare Network, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - Geisinger Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Main Line Health, Wynnewood, Pennsylvania
  - Cardiology Consultants of Philadelphia | Yardley, Yardley, Pennsylvania
  - Lifespan | The Miriam Hospital - Cardiovascular Research, Providence, Rhode Island
  - AnMed Clinical Research, Anderson, South Carolina
  - Medical University of South Carolina - Cardiology, Charleston, South Carolina
  - Piedmont Research Partners LLC, Fort Mill, South Carolina
  - Accellacare | Mt. Pleasant, SC, Ladson, South Carolina
  - Carolina Heart Specialists | Lancaster, SC, Lancaster, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Holston Medical Group - Bristol, Bristol, Tennessee
  - Erlanger Health, Inc., Chattanooga, Tennessee
  - Stern Cardiovascular Center, Germantown, Tennessee
  - Apex Research Foundation, LLC. | Jackson, TN, Jackson, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cardiovascular Research of Knoxville, Powell, Tennessee
  - PharmaTex Research, LLC, Amarillo, Texas
  - Southwest Family Medicine Associates | Dallas, TX, Dallas, Texas
  - Prime Revival Reserach Institute, LLC | Denton, TX, Denton, Texas
  - David Turbay MD PLLC, El Paso, Texas
  - Texas Health Research & Education Institute, Fort Worth, Texas
  - Texas Health Physicians Group - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - TCR Institute, Kingwood, Texas
  - North Dallas Research Associate | McKinney, TX, McKinney, Texas
  - North Texas Research Associates, McKinney, Texas
  - Styde Research LLC | Plano, TX, Plano, Texas
  - South Texas Cardiovascular Consultants, PLLC, San Antonio, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Mt. Olympus Medical Research, Sugar Land, Texas
  - Northwest Houston Clinical Research, PLLC - Houston Heart Center | Tomball, TX, Tomball, Texas
  - Tyler Cardiovascular Consultants | Tyler, TX, Tyler, Texas
  - CHRISTUS Trinity | Mother Frances Louis and Peaches Owen Heart Hospital - Electrophysiology Clinic, Tyler, Texas
  - Intermountain Healthcare | Cardiovascular Research Department, Murray, Utah
  - Inova Fairfax Hospital - Fairfax, Fairfax, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Carient Heart and Vascular, Manassas, Virginia
  - York Clinical Research, LLC | Norfolk, VA, Norfolk, Virginia
  - Hunter Holmes McGuire Veterans Affairs Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Sound Medical Research | Sound Medical Research of Port Orchard, Port Orchard, Washington
  - Confluence Health, Wenatchee, Washington
- Argentina (17):
  - Instituto de Investigaciones Clinicas Bahia Blanca | Bahia Blanca, Argentina, Bahía Blanca, Buenos Aires
  - Centro de Investigación y Prevención Cardiovascular, General Arenales, Buenos Aires
  - Hospital Italiano de La Plata | Clinical Research Department, La Plata, Buenos Aires
  - Centro de Investigaciones Medicas Lanus | Buenos Aires, Argentina, Lanús, Buenos Aires
  - Instituto de Investigaciones Clinicas de Mar del Plata | Mar del Plata, Argentina, Mar del Plata, Buenos Aires
  - CardioAlem Investigaciones | San Isidro, Argentina, San Isidro, Buenos Aires
  - Instituto de Investigaciones Clínicas (IIC) San Nicolas | San Nicolas de los Arroyos, Argentina, San Nicolás de los Arroyos, Buenos Aires
  - Centro de Investigaciones Medicas Temperley | Buenos Aires, Argentina, Temperley, Buenos Aires
  - Instituto De Investigaciones Clinicas Zarate | Zarate, Argentina, Zárate, Buenos Aires
  - Centro de Investigaciones Metabolicas | Ciudad de Autonoma de Buenos Aires, Argentina, Buenos Aires, Ciudad Auton. de Buenos Aires
  - CEDIC Centro de Investigación Clínica | Buenos Aires, Argentina, CABA, Ciudad Auton. de Buenos Aires
  - Centro de Especialidades Medicas (Cemedic) | Cardiology Department, Villa Luro, Ciudad Auton. de Buenos Aires
  - Consultorios Integrados Rosario | Instituto Medico de la Fundacion de Estudios Clinicos, Rosario, Santa Fe Province
  - Laboratorio de Hemostasia y Trombosis | Rosario, AR, Rosario, Santa Fe Province
  - Investigaciones Clinicas Tucuman | San Miguel de Tucuman, Argentina, San Miguel de Tucumán, Tucumán Province
  - Instituto de Cardiologia de Corrientes Juana F. Cabral | Corrientes, Argentina, Corrientes
  - Centro de Investigaciones Clinicas del Litoral | Santa Fe, Argentina, Santa Fe
- Australia (30):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Blacktown Hospital, Blacktownn, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - South Western Sydney Local Health District | Liverpool Hospital - Stroke and Neurovascular Department, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Illawarra Shoalhaven Local Health District, Wollongong, New South Wales
  - Advara HealthCare Wesley, Auchenflower, Queensland
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane & Women's Hospital, Brisbane, Queensland
  - The Prince Charles Hospital, Herston, Queensland
  - Redcliffe District Hospital, Redcliffe, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Core Research Group Pty Ltd. | Brisbane, Australia, Taringa QLD, Queensland
  - Nightingale Research, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Advara HealthCare Leabrook, Leabrook, South Australia
  - Queen Elizabeth Hospital AUS, Woodville South, South Australia
  - Grampians Health Ballarat, Ballarat, Victoria
  - Eastern Health, Box Hill, Victoria
  - Barwon Health, Geelong, Victoria
  - Baker Heart and Diabetes Institute, Hoppers Crossing, Victoria
  - Cabrini Malvern, Malvern, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Advara HeartCare Melbourne, Ringwood, Victoria
  - The Avenue Cardiovascular Centre, St Kilda East, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Advara HealthCare Joondalup, Perth, Western Australia
  - Nepean Hospital, Kingswood
- Austria (16):
  - Klinikum Klagenfurt | Innere Medizin und Kardiologie, Klagenfurt, Carinthia
  - Landesklinikum Mistelbach|Kardiologie u. Internistische Med, Mistelbach, Lower Austria
  - UK St. Poelten | Innere Med III, Sankt Pölten, Lower Austria
  - MedUni Graz | Kardiologie, Graz, Styria
  - Landeskrankenhaus Hall | Abteilung fuer Innere Medizin, Hall in Tirol, Tyrol
  - MedUni Innsbruck | Kardiologie und Angiologie, Innsbruck, Tyrol
  - Krankenhaus St. Josef Braunau | Innere Medizin I, Braunau am Inn, Upper Austria
  - Elisabethinen Linz | Kardiologie, Angiologie & Intensiv Med, Linz, Upper Austria
  - Kepler UK Linz | Kardiologie & Intensivmedizin Campus III, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen | Innere Medizin II, Wels, Upper Austria
  - MedUni Wien | Innere Medizin II, Kardiologie, Vienna, Vienna
  - Klinik Floridsdorf | Herz-, Gefaess- u. Kardio Ambulaz, Vienna, Vienna
  - LKH Feldkirch | Innere Medizin I mit Kardiologie, Feldkirch, Vorarlberg
  - Uniklinikum Salzburg|Innere Medizin II, Kardiologie, Salzburg
  - Hanusch Krankenhaus | 2. Medizinische Abteilung, Vienna
  - Imed19-privat, Vienna
- Belgium (23):
  - Imelda Vzw | Study Cardiology, Bonheiden, Antwerpen
  - Antwerp University Hospital | Cardiology Department, Edegem, Antwerpen
  - GZA Ziekenhuizen | Saint Augustine Campus - Cardiology Department, Wilrijk, Antwerpen
  - CHC MontLégia Neurology Department, Liège, Liège
  - University Hospital Louvain Namur | Godinne - Cardiology Department, Yvoir, Namur
  - AZ St-Lucas Campus St-Lucas - Cardiology, Ghent, Oost-Vlaanderen
  - Maria Middelares General Hospital | Cardiology Department, Ghent, Oost-Vlaanderen
  - UZ Leuven Gasthuisberg, Leuven, Vlaams Brabant
  - Groeninge Algemeen Ziekenhuis | Campus Kennedylaan - Cardiology Departement, Kortrijk, West-Vlaanderen
  - Algemeen Stedelijk Ziekenhuis Campus Aalst, Aalst
  - OL Vrouwziekenhuis - Campus Aalst, Aalst
  - ZNA Middelheim, Antwerp
  - Algemeen Ziekenhuis Klina | Cardiology Department, Brasschaat
  - AZ Sint-Jan Brugge-Oostende | Sint-Jan - Cardiology, Bruges
  - CU Saint-Luc/UZ St-Luc, Bruxelles - Brussel
  - AZ Sint Blasius, Cardiology, Dendermonde, Dendermonde
  - AZ Sint-Maarten, Duffel
  - Ziekenhuis Oost-Limburg | Genk, Sint-Jan campus - Cardiology Department, Genk
  - Grand Hôpital de Charleroi, Gilly
  - Jessa Ziekenhuis, Hasselt
  - Citadelle Hospital | Cardiology Department, Liège
  - AZ Delta | Clinical Trial Center - Cardiology, Roeselare
  - Vitaz | Sint-Niklaas Hospital - Cardiology Department, Sint-Niklaas
- Brazil (26):
  - Hospital Cardio Pulmonar | Salvador, Brazil, Salvador, Estado de Bahia
  - Hospital das Clinicas da Universidade Federal de Goias | Centro de Pesquisa em Cardiologia, Goiânia, Goiás
  - Cardresearch Cardiologia Assistencial e de Pesquisa | Belo Horizonte, Brazil, Belo Horizonte, Minas Gerais
  - Hospital Maternidade e Pronto Socorro Santa Lucia | Hospital do Coracao - Research Center, Poços de Caldas, Minas Gerais
  - Quanta Diagnostico Por Imagem | Research and Innovation Department, Curitiba, Paraná
  - Nucleo de Pesquisa Clinica | Curitiba, Brazil, Curitiba, Paraná
  - Centro Medico Sao Francisco | Curitiba, Brazil, Curitiba, Paraná
  - Sociedade Hospitalar Angelina Caron | Departamento de Ensino e Pesquisa, Paraná, Paraná
  - Irmandade da Santa Casa de Misericordia de Porto Alegre | Hospital Sao Francisco - Centro Medico Pesquisa Clinica Cardiologia, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre | Clinical Research Center - Surgery Research Center, Porto Alegre, Rio Grande do Sul
  - FZ Pesquisa e Servicos em Cardiologia | Porto Alegre, Brazil, Porto Alegre, Rio Grande do Sul
  - CardioBlu | Unidade Sabin, Blumenau, Santa Catarina
  - Centro de Pesquisa Clinica do Coração | Aracaju, Brasil, Aracaju, Sergipe
  - UNESP Faculdade de Medicina de Botucatu | UPECLIN, Botucatu, São Paulo
  - Campinas Clinical Research Institute (IPECC) | Campinas, Brazil, Campinas, São Paulo
  - Instituto do Coração de Marilia | Marilia, Brasil, Marília, São Paulo
  - Hospital e Maternidade Christovao da Gama | Santo Andre Medical Centre - Cardiology Department, Santo André, São Paulo
  - Hospital de Base | Integrated Research Center, São José do Rio Preto, São Paulo
  - Irmandade da Santa Casa de Misericordia de Sao Paulo | Hospital Central - Cardiology Department, São Paulo, São Paulo
  - Hospital Samaritano Paulista | Clinical Research Department, São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia | Divisao de Pesquisa, São Paulo, São Paulo
  - Hospital e Maternidade Sao Luiz, São Paulo, São Paulo
  - Hospital PUC-Campinas | Centro de Pesquisa Clínica Sao Lucas, São Paulo, São Paulo
  - Eurolatino Pesquisas Medicas | Uberlandia, MG, Minas Gerais
  - Hospital Sao Lucas Copacabana | Clinical Research Department, Rio de Janeiro
  - Hospital Alemao Oswaldo Cruz | Centro Internacional de Pesquisa, São Paulo
- Bulgaria (23):
  - Multiprofile Hospital for Active Treatment Puls | Clinical Trial Center, Blagoevgrad
  - Multidisciplinary Hospital for Active Treatment Heart and Brain Burgas | Cardiology Department, Burgas
  - Medical Center Avitsena Kardzhali | Cardiology Clinic, Kardzhali
  - SHATC Sveti Georgi - Pernik | Pernik, Bulgaria, Pernik
  - Medical centre Hipokrat - N EOOD, Plovdiv
  - Multiprofile Hospital for Active Treatment Medline | Cardiology Department, Plovdiv
  - Multiprofile Hospital for Active Treatment Sveta Karidad | Cardiology Department, Plovdiv
  - Medical Center Rusemed EOOD | Ruse, Bulgaria, Rousse
  - Multiprofile Hospital for Active Treatment | Shumen - First Department of Internal Medicine, Shumen
  - General Hospital Silistra | Department of Cardiology, Structure for Interventional Cardiology, Silistra
  - Cardiohelp Medical Centre | Sofia, Bulgaria, Sofia
  - Diagnostic Consultative Center Ascendent | Sofia, Bulgaria, Sofia
  - Second Medical Center Sofia EOOD, Sofia
  - Multiprofile Hospital for Active Treatment Knyaginya Klementina Sofia EAD | Cardiology Department, Sofia
  - Multiprofile Hospital for Active Treatment National Cardiology Hospital | Cardiology Department, Sofia
  - University Hospital for Active Treatment Tsaritsa Joanna - ISUL | Cardiology Clinic, Sofia
  - The University General Hospital for Active Care and Emergency Medicine Pirogov | Cardiology Department, Sofia
  - Diagnostic-Consultative Center XX | Cardiology Department, Sofia
  - Multiprofile Hospital for Active Treatment Sveta Sofia | Internal Diseases Department, Sofia
  - Multiprofile Hospital for Active Treatment Trakiya Park | Cardiology Department, Stara Zagora
  - Medical Center Zara-Med EOOD | Cardiology Department, Stara Zagora
  - NOVA Clinic Medical Center | Varna, BG, Varna
  - Multiprofile Hospital for Active Treatment Dr. Stefan Cherkezov | Cardiology Department, Veliko Tarnovo
- Canada (40):
  - Edmonton Cardiology Consultants, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Interior Health - Royal Inland Hospital, Kamloops, British Columbia
  - Fraser Clinical Trials, Inc., New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - G.A. Research Associates, Ltd., Moncton, New Brunswick
  - Memorial University of Newfoundland, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Cambridge Cardiac Care Center, Cambridge, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - Hamilton Med.Research Group - DCT, Hamilton, Ontario
  - Hamilton Medical Research Group, Hamilton, Ontario
  - St. Joseph's Healthcare - Hamilton, Hamilton, Ontario
  - Milestone Research, London, Ontario
  - London Health Sciences Centre | University Hospital - London Heart Rhythm Program - Cardiology, London, Ontario
  - Oakville Cardiovascular Research, Oakville, Ontario
  - Dr. James Cha, Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Heart Health Institute, Scarborough Village, Ontario
  - Niagara Health - St. Catharines Site, St. Catharines, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital UHN, Toronto, Ontario
  - Women's College Hospital | WCH Main Site - Women's College Research Institute - Cardiology Department, Toronto, Ontario
  - Dr. Louis Yao, York, Ontario
  - Viacar Recherches Cliniques Inc., Brossard, Quebec
  - CIUSSS Saguenay Lac-St-Jean, Chicoutimi, Quebec
  - Centre intégré de santé et de services sociaux de Laval, Hôp, Laval, Quebec
  - Centricity Research Mirabel Multispecialty, Mirabel, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - CHUM - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - McGill University Health Centre - Glen Site, Montreal, Quebec
  - CIUSSS NÎM Hôpital Sacré-Coeur, Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
  - CIUSSS de l'Estrie-CHUS, Hopital Fleurimont, Sherbrooke, Quebec
  - CISSSL - Hopital Pierre-Le Gardeur, Terrebonne, Quebec
  - Diex Research Trois-Rivières Inc., Trois-Rivières, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Q, Québec
- China (88):
  - The 1st Affiliated Hospital Fujian Medical University, Fuzhou, Fujian
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangzhou First People Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of TCM, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - The 2nd Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Hainan Provincial People's Hospital, Haikou, Hainan
  - Hainan Third People's Hospital (Province Nongken Sanya Hopt), Sanya, Hainan
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - The First Hospital of Hebei Medical Univesity, Shijiazhuang, Hebei
  - The First affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The 4th Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - 1st Affiliated Hospital of Henan Science and Technology Univ, Luoyang, Henan
  - Luoyang Third People's Hospital, Luoyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - The Central Hospital of Wuhan, Tongji Medl Collg Huazhong..., Wuhan, Hubei
  - Union Hospt Tongji Medical Colleg. Huazhong univ. Scien&Tech, Wuhan, Hubei
  - Puai Hospital,Tongji Medical College, Huazhong Univ Sci&Tech, Wuhan, Hubei
  - Renmin Hosp., Wuhan Univ., Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Hospital of Changsha, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - Huai'an First People's Hospital, Nanjing Medical University, Huai'an, Jiangsu
  - Affiliated Hospital of Jiangsu University, JiangSu, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical university, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Affiliated Hospital of Yangzhou University (Yangzhou First People's Hospital), Yangzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - Jiangxi PingXiang people's Hospital, Pingxiang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Tonghua Central Hospital, Tonghua, Jilin
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Panjin Liaohe Oilfield Gem Flower Hospital, Panjin, Liaoning
  - Yinchuan No.1 People's Hospital, Yinchuan, Ningxia
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - Yan'an University Xianyang Hospital, Xianyang, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - The 2nd Affiliated Hospital of Shandong University, Jinan, Shandong
  - Qilu Hosp., Shandong Univ., Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Jining No.1 People's Hospital, Jining, Shandong
  - Taian City Central Hospital, Taian, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Shanxi Candiovascular Hospital, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shaanxi Provincial People's Hospital, Xi’an, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - SichuanAcademyofMedicalSciences&SichuanProvincialPeople'sHos, Chengdu, Sichuan
  - People's Hospital of Deyang City, Deyang, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The 1st Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Affiliated Hangzhou First People's Hospital, Zhejiang Univ, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Hwa Mei Hospital, University of Chinese Academy Sciences, Ningbo, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Beijing Tongren Hospital, Capital Medical University (West), Beijing
  - Peking Union Medical College Hospital CAMS, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Zhongshan Hospital, Fudan University, Shanghai
  - Huashan Hospital, Fudan University, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanghai Putuo District Central Hospital, Shanghai
  - Tianjin People's Hospital, Tianjin
  - Teda International Cardiovascular Hospital, Tianjin
- Czechia (20):
  - Benedor s.r.o., Ostrava - Poruba, Moravskoslezský kraj
  - Cevni Kulatak, Prague, Prague
  - Cardio Research s.r.o., Zlín, Zlín
  - Kardiologicka ambulance Brno s.r.o., Brno
  - Fakultni nemocnice Brno, Brno
  - Vojenska nemocnice Brno, Brno
  - Amkardia s.r.o., Brno
  - Kardiologicka ambulance Cormedico, Bruntál
  - Nemocnice Ceske Budejovice, a.s. Department of kardiologie, České Budějovice
  - Mrozek kardiologie, Frýdek-Místek
  - MATMED s.r.o., Hodonín
  - Krajska Nemocnice Liberec, Liberec
  - Fakultni Nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Plzen, Pilsen
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Institut Klinicke a Experimentalni Mediciny, Prague
  - Fakultni nemocnice v Motole, Prague
  - Medicon Poliklinika Holesovice, Prague
  - Nemocnice Slany, Slaný
  - MUDr. Michalik s.r.o., Zábřeh nad Odrou
- Denmark (16):
  - Region Nordjylland | Aalborg University Hospital - Cardiology Department, Aalborg
  - Region Midtjylland | Aarhus University Hospital - Heart Diseases - Clinical Research, Århus N
  - Capital Region | Amager Hospital - Cardiology Outpatient Clinic, Copenhagen
  - Sydvestjysk Sygehus Esbjerg | Kardiologisk Forskningsenhed, Esbjerg
  - Capital Region | Frederiksberg Hospital - Department of Cardiology Research, Frederiksberg
  - Capital Region | Gentofte Hospital - Cardiology Research, Hellerup
  - Capital Region | Herlev Hospital - Department of Heart Disease, Herlev
  - Region Midtjylland | Regionshospitalet Godstrup - Clinic for Heart Research, Herning
  - Capital Region | Nordsjaellands Hospital - Hillerod - Cardiology Department, Hilleroed
  - Region Nordjylland | Hjoerring - Cardiology Department, Hjørring
  - Region Sjælland | Holbaek Sygehus - Cardiology department, Holbæk
  - Capital Region | Hvidovre Hospital - Department of Cardiology, Hvidovre
  - Sygehus Lillebaelt | Kolding Sygehus - Medicinske Sygdomme, Kolding
  - Sjællands Universitetshospital Roskilde - Hormon og stofskiftesygdomme, Roskilde
  - Odense University Hospital | Svendborg Hospital - Cardiovascular Research Unit, Svendborg
  - Region Midtjylland | Viborg Regional Hospital - Cardiology - Heart Research, Viborg
- Estonia (8):
  - Rapla Family Doctors Centre, Rapla
  - Dr Signe Alliksoo Family Doctors Practice, Tallinn
  - East Tallinn Central Hospital, Tallinn
  - Pirita Family Doctors Centre, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Office of Arvo Rosenthal, Tallinn
  - West Tallinn Central hospital, Tallinn
  - Tartu University Hospital, Tartu
- Finland (10):
  - HUS Jorvin sairaala, Espoo
  - StudyCor Oy, Jyväskylä
  - Keski-Pohjanmaan keskussairaala, Kokkola
  - Health Step Finland Oy, Kuopio
  - Kuopion yliopistollinen sairaala, Kuopio
  - Päijät-Hämeen keskussairaala, Lahti
  - Oulun yliopistollinen sairaala, Oulu
  - Tays Sydänsairaala, Tampere
  - Terveystalo Pulssi, Turku
  - Turun yliopistollinen keskussairaala, Turku
- France (33):
  - Centre Hospitalier Universitaire - Angers, Angers
  - Centre Hospitalier Intercommunal de la Côte Basque-Bayonne, Bayonne
  - Hopital Charles Nicolle Chu Rouen, Bois-Guillaume
  - Hôpital La Cavale Blanche - CHU de Brest, Brest
  - Hôpital Louis Pradel - Bron, Bron
  - CHU de Caen - Hôpital Côte de Nacre, Caen
  - Hôpital Trousseau - Tours, Chambray-lès-Tours
  - Centre Hospitalier - Cholet, Cholet
  - Hôpital Henri Mondor, Créteil
  - CHU GRENOBLE - Hopital Michallon, Grenoble
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Centre Hospitalier Louis Pasteur, Le Coudray
  - Centre Hospitalier du Docteur Schnaffer - Lens, Lens
  - Hôpital Dupuytren, Limoges
  - Hôpital Arnaud de Villeneuve - Montpellier, Montpellier
  - Hôpital Guillaume et René Laennec - Nantes, Nantes
  - Nouvelles Cliniques Nantaises - Nantes, Nantes
  - Hôpital Pasteur - Nice, Nice
  - Hopital Carémeau - Nîmes, Nîmes
  - Institut Mutualiste Montsouris, Paris
  - Hôpital de la Pitié-Salpétrière, Paris
  - Hopital Européen Georges Pompidou - Paris, Paris
  - Hôpital Cardiologique - Pessac, Pessac
  - CHU Rennes, H Pontchaillou, Cardiologie, Rennes
  - Centre Hospitalier Régional - Saint Brieuc, Saint-Brieuc
  - Centre de Cardiologie Nord - Saint Denis, Saint-Denis
  - Hôpital Civil - Strasbourg, Strasbourg
  - CHI Toulon - H La Seyne - Cardiologie, Toulon
  - Hôpital de Rangueil - Toulouse, Toulouse
  - Clinique Pasteur - Toulouse, Toulouse
  - Centre Hospitalier Gustave Dron - Tourcoing, Tourcoing
  - Centre Hospitalier - Valenciennes Cedex, Valenciennes
  - Centre Hospitalier Universitaire de Nancy, Vandœuvre-lès-Nancy
- Germany (29):
  - Universitaets Herzzentrum Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - Uni-Klinikum Heidelberg | Kardiologie Angiologie Pneumologie, Heidelberg, Baden-Wurttemberg
  - MEDICLIN Herzzentrum Lahr|Kardiologie, Lahr, Baden-Wurttemberg
  - Cardio Centrum Ludwigsburg, Ludwigsburg, Baden-Wurttemberg
  - Hegau-Bodensee-Klinikum Singen|I. Medizinische Klinik, Singen, Baden-Wurttemberg
  - Klinikum Fulda gAG|Medizinische Klinik I, Fulda, Hesse
  - Medizinische Hochschule Hannover|Kardiologie und Angiologie, Hanover, Lower Saxony
  - UniKlinikum Aachen|Kardio, Angio, Intensivmedizin, Aachen, North Rhine-Westphalia
  - St. Vinzenz-Hospital|Innere Medizin III, Kardiologie, Cologne, North Rhine-Westphalia
  - St.Johannes-Hospital|Klinik fuer Innere Medizin I, Dortmund, North Rhine-Westphalia
  - Ev. Krankenhaus Hagen-Haspe|Kardiologie und Rhythmologie, Hagen, North Rhine-Westphalia
  - Klinikum Lüdenscheid - Märkische Kliniken GmbH, Lüdenscheid, North Rhine-Westphalia
  - Kliniken Maria Hilf GmbH, Mönchengladbach, North Rhine-Westphalia
  - Sana-Klinikum Remscheid|Kardio, Angio, Pneumo u. Intensivmed, Remscheid, North Rhine-Westphalia
  - Josephs-Hospital|Kardiologie, Rhythmologie und Angiologie, Warendorf, North Rhine-Westphalia
  - Forschungszentrum Ruhr KliFoCenter GmbH, Witten, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
  - Klinikum Worms gGmbH|Kardiologie und Angiologie, Worms, Rhineland-Palatinate
  - Siteworks Pruefzentrum Voelklingen, Völklingen, Saarland
  - Klinische Forschung Dresden | Dresden, Germany, Dresden, Saxony
  - Krankenhaus Dresden-Friedrichstadt, Dresden, Saxony
  - Praxisklinik Herz und Gefaesse|Kardiologische Ambulanz, Dresden, Saxony
  - Uniklinik Leipzig / Kardiologie, Leipzig, Saxony
  - Praxis Hr. Dr. med. Jens Taggeselle, Markkleeberg, Saxony
  - Kardiologische Praxis Hr. Dr. A. Al-Zoebi, Wermsdorf, Saxony
  - Uniklinik Jena / Kardiologie, Jena, Thuringia
  - Uniklinikum Hamburg-Eppendorf|Klinik für Kardiologie, Hamburg
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Cardiologicum Hamburg, Hamburg
- Greece (21):
  - KAT General Hospital of Athens, Kifissia, Attica
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - General Hospital of Athens "Evangelismos", Athens
  - HIPPOKRATION General Hospital of Athens, Athens
  - Naval Hospital of Athens, Athens
  - G. GENNIMATAS General State Hospital of Athens, Athens
  - LAIKO General Hospital of Athens, Athens
  - General Hospital of Athens "ALEXANDRA", Athens
  - University General Hospital of Athens "ATTIKON", Chaïdári
  - Thriassio General Hospital of Elefsina, Elefsina
  - University General Hospital of Heraklion, Heraklion
  - Univ. General Hospital of Ioannina, Ioannina
  - University General Hospital of Ioannina, Ioannina
  - Univ. General Hospital of Larissa, Larissa
  - University General Hospital of Larissa, Larissa
  - MITERA Hospital, Marousi
  - Konstantopoulio General Hospital of Nea Ionia - AGIA OLGA, Nea Ionia
  - University General Hospital of Patra, Pátrai
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
  - Hippokration General Hospital of Thessaloniki, Thessaloniki
  - General Hospital ASKLEPIEIO VOULAS, Voula
- Hungary (22):
  - Cardiomobile Egeszsegugyi Szolgaltato Kft., Balatonfüred
  - Budapesti Jahn Ferenc Del-pesti Korhaz es Rendelointezet, Budapest
  - Semmelweis University, Budapest
  - Budapesti Uzsoki Utcai Korhaz, Budapest
  - Belinus Bt., Debrecen
  - Kardio Egeszseghaz - Dr Amer Sayour Egyeni Vallakozo, Győr
  - Trial Pharma Kft. Gyula, Gyula
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Komaromi Selye Janos Korhaz, Komárom
  - Borsod-Abauj-Zemplen Varmegyei Korhaz es Egyetemi Oktatokorhaz, Miskolc
  - TaNa Med Kft., Mosonmagyaróvár
  - Nagykanizsai Kanizsai Dorottya Korhaz, Nagykanizsa
  - Medifarma-98 Egeszsegugyi, Kereskedelmi es Szolgaltato Kft., Nyíregyháza
  - Borbanya Praxis Bt., Nyíregyháza
  - Dr. Laszlo Elek Korhaz es Rendelointezet, Oroshaza, Orosháza
  - Dr. Nagy Laszlo Egyeni Egeszsegugyi Vallalkozo, Orosháza
  - Coromed Smo Kft, Pécs
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Tolna Varmegyei Balassa Janos Korhaz, Szekszárd
  - Complex Rendelo Med Zrt., Székesfehérvár
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz, Szombathely
  - Belvarosi Egeszseghaz Kft., Zalaegerszeg
- India (4):
  - Lisie Hospital, Kochi, Kerala
  - Vijan Cardiac & Critical Care Centre, Nashik, Maharashtra
  - Asian Institute of Gastroenterology (AIG Hospital), Hyderabad
  - King Edward Memorial (KEM) Hospital - Pune, Pune
- Israel (23):
  - HaEmek Medical Center | Internal Medicine C Department - Research Unit, Afula
  - Samson Assuta Ashdod University Hospital | Cardiology Department, Ashdod
  - Barzilai Ashkelon University Medical Center | Cardiology Department, Ashkelon
  - Clalit Health | Soroka Medical Center - Cardiology Department, Beersheba
  - Clalit Health | Soroka Medical Center - Internal Medicine Department, Beersheba
  - Assuta Hospital Be'er Sheva | Heart Institute - Clinics, Beersheba
  - Hillel Yaffe Medical Center | Cardiology Department, Hadera
  - Rambam Health Care Campus | Cardiology Department - Cardiology Research Unit, Haifa
  - Bnai Zion Medical Center | Cardiology Department, Haifa
  - Carmel Medical Center | Cardiology Department - Cardiac Catheterization Unit, Haifa
  - Edith Wolfson Medical Center | Internal Medicine Department, Holon
  - Shaare Zedek Medical Center | The Jesselson Integrated Heart Center - Cardiology Department, Jerusalem
  - Clalit Health | Meir Medical Center - Division of Cardiology - Electrophysiology and Arrhythmias Unit, Jerusalem
  - Hadassah Hebrew University Hospital Ein Kerem, Jerusalem
  - Poria Medical Center | Cardiovascular Department, Lower Galilee
  - Galilee Medical Center | Cardiology Department, Nahariya
  - Rabin Medical Center | Beilinson Hospital - Internal Medicine C Department, Petah Tikva
  - Rabin Medical Center | Clinical Trials Unit - Cardiology Department, Petah Tikva
  - Kaplan Medical Center | Cardiology Department - Heart Institute Research, Rehovot
  - Shamir Medical Center | Cardiology Department, Rishon LeZiyyon
  - Ziv Medical Center | Cardiology Department, Safed
  - Tel Aviv Sourasky Medical Center | Ichilov General Hospital - Cardiology Department, Tel Aviv
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (29):
  - ASL2 Lanciano-Vasto-Chieti, Chieti, Abruzzo
  - Ente Ecclesiastico Ospedale Generale Regionale Miulli, Bari, Apulia
  - A.O.U. Ospedali Riuniti Foggia, Foggia, Apulia
  - A.O Sant'Anna-San Sebastiano, Caserta, Campania
  - A.O.U. Policlinico Federico II Napoli, Naples, Campania
  - A.O.R.N. Ospedali dei Colli (Monaldi-Cotugno-CTO), Napoli, Campania
  - Azienda Unita Sanitaria Locale Di Bologna_Ospedale Maggiore Pizzardi - Cardiologia, Bologna, Emilia-Romagna
  - A.O.U. di Ferrara, Ferrara, Emilia-Romagna
  - A.O.U. di Modena - Policlinico, Modena, Emilia-Romagna
  - A.O.U. di Parma, Parma, Emilia-Romagna
  - Asl Roma 2, Rome, Lazio
  - A.O.U. Policlinico Umberto I, Rome, Lazio
  - ASST Papa Giovanni XXIII, Bergamo, Lombardy
  - ASST del Garda, Brescia, Lombardy
  - Ospedale San Raffaele s.r.l. - Cardiologia Clinica, Milan, Lombardy
  - IRCCS Centro Cardiologico Monzino, Milan, Lombardy
  - Humanitas Mirasole S.p.A. - Centro Trombosi e Malattie Emorragiche, Rozzano, Lombardy
  - ASST Sette Laghi, Varese, Lombardy
  - A.O.U. Maggiore della Carità, Novara, Piedmont
  - A.O.U. Policlinico G. Martino, Messina, Sicily
  - A.O.U. Ospedali Riuniti "Umberto I - G.M.Lancisi - G.Salesi", Ancona, The Marches
  - ASUR Marche - Area Vasta 5, Ascoli Piceno, The Marches
  - AUSL Toscana Sud-Est, Arezzo, Tuscany
  - A.O.U. Careggi, Florence, Tuscany
  - A.O.U. Pisana, Pisa, Tuscany
  - A.O. di Perugia, Perugia, Umbria
  - A.O.U. di Padova, Padua, Veneto
  - ULSS2 Marca Trevigiana, Treviso, Veneto
  - ULSS3 Serenissima, Venezia, Veneto
- Japan (119):
  - Kasugai Municipal Hospital, Kasugai, Aichi-ken
  - Japan Community Healthcare. Organization Chukyo Hospital, Nagoya, Aichi-ken
  - Japanese RedCross Aichi Medical Center Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Japan Culture and Welfare Federation of Agricultural Cooperatives | Toyota Kosei Hospital, Toyota, Aichi-ken
  - Chiba Tokushukai Hospital | Clinical Trial Center, Funabashi, Chiba
  - Nippon Medical School Chiba Hokusoh Hospital | Clinical Trial Office, Inzai, Chiba
  - Kimitsu Chuo Hospital, Kisarazu, Chiba
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Matsuyama Shimin Hospital, Matsuyama, Ehime
  - Munakata Suikokai General Hospital | Cardiology Department, Fukutsu, Fukuoka
  - Nakamura Cardiovascular Clinic, Itoshima, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Steel Memorial Yawata Hospital, Kitakyushu, Fukuoka
  - Go Neurosurgical Clinic, Nakagawa, Fukuoka
  - Onga Nakama Medical Association Onga Hospital, Onga-gun, Fukuoka
  - Fukuoka Shinmizumaki Hospital | Clinical Trial Management Office, Tateyashiki, Mizumakimachi, on, Fukuoka
  - Yanagawa Hospital, Yanagawa, Fukuoka
  - Japan Culture and Welfare Federation of Agricultural Cooperatives | ShirakawaKosei General Hospital, Shirakawa, Fukushima
  - National Hospital Organization Takasaki General Medical Center, Takasaki, Gunma
  - Mazda Motor Corporation Mazda Hospital, Aki-gun, Hiroshima
  - Asahikawa City Hospital, Asahikawa, Hokkaido
  - Hakodate National Hospital, Hakodate, Hokkaido
  - Hakodate Municipal Hospital, Hakodate, Hokkaido
  - Matsuda Cardiovascular clinic, Sapporo, Hokkaido
  - Mita Internist and Cardiology Clinic | Hokkaido, Japan, Sapporo, Hokkaido
  - Teine Keijinkai Hospital, Sapporo, Hokkaido
  - Hanaoka Seishu Memorial Hospital, Sapporo, Hokkaido
  - Miyanosawa Clinic of Internal Medicine and Cardiology, Sapporo, Hokkaido
  - Miyanomori Memorial Hospital, Sapporo, Hokkaido
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Oji General Hospital, Tomakomai, Hokkaido
  - Tomakomai City Hospital, Tomakomai, Hokkaido
  - Akashi Medical Center | Hyogo, Japan, Akashi, Hyōgo
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki, Hyōgo
  - Hyogo Prefectural HarimaHimeji General Medical Center, Himeji, Hyōgo
  - The Veritas Hospital, Kawanishi, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Higashi Takarazuka Satoh Hospital, Takarazuka, Hyōgo
  - National hospital Organization Mito Medical Center, Higashiibaraki, Ibaraki
  - Ibaraki Prefectural Central Hospital, Kasama, Ibaraki
  - Mito Saiseikai General Hospital, Mito, Ibaraki
  - JA Toride Medical Center, Toride, Ibaraki
  - Tsuchiura Kyodo General Hospital, Tsuchiura, Ibaraki
  - Public Central Hospital of Matto Ishikawa | Clinical Trial Management Office, Hakusan, Ishikawa-ken
  - Kanazawa Medical University Hospital, Kahoku-gun, Ishikawa-ken
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - National Hospital Organization Kanazawa Medical Center | Clinical Trial Management Office, Kanazawa, Ishikawa-ken
  - Komatsu Municipal Hospital, Komatsu, Ishikawa-ken
  - Iwate Prefectural Central Hospital, Morioka, Iwate
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Mitoyo General Hospital | Kagawa, Japan, Toyohama-Cho,Kanonji-City, Kagawa-ken
  - Oosumikanoya Hospital, Kanoya, Kagoshima-ken
  - Fujisawa City Hospital, Fujisawa, Kanagawa
  - Hayama Heart Center | Clinical Trial Center, Miura-gun, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Yokohama Sakae Kyosai Hospital, Yokohama, Kanagawa
  - Japan Culture and Welfare Federation of Agricultural Cooperatives | Suzuka Chuo General Hospital, Suzuka-shi, Mie-ken
  - Sendai Cardiovascular Center, Sendai, Miyagi
  - Tohoku Medical and Pharmaceutical University Hospital | Center for Clinical Research Promotion and Development, Sendai, Miyagi
  - Japan Red Cross Society Azumino Hospital, Azumino, Nagano
  - Iida Hospital, Iida, Nagano
  - North Alps Medical Center Azumi Hospital, Kitaazumi-gun, Nagano
  - Asama Nanroku Komoro Medical Center | Komoro, Japan, Komoro, Nagano
  - Japan Culture and Welfare Federation of Agricultural Cooperatives | Hokushin General Hospital, Nakano, Nagano
  - Japanese Red Cross Society Suwa Hospital, Suwa, Nagano
  - R.I.A.C Naha City Hospital, Naha, Okinawa
  - Urasoe General Hospital | Clinical Research Support Center, Urasoe, Okinawa
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Osaka Saiseikai Senri Hospital, Suita, Osaka
  - Sakurabashi Watanabe Future Medical Hospital | Department of Cardiology, Umeda Kita-Ku, Osaka-shi, Osaka
  - Yao Tokushukai General Hospital | Clinical Research Center, Yao, Osaka
  - Ageo Central General Hospital, Ageo, Saitama
  - Kawaguchi Cardiovascular and Respiratory Hospital, Kawaguchi, Saitama
  - Omihachiman Community Medical Center, Ōmihachiman, Shiga
  - National Hospital Organization Hamada Medical Center, Hamada, Shimane
  - Dokkyo Medical University Hospital, Shimotsuga-gun, Tochigi
  - Tokyo Medical and Dental University Hospital, Bunkyo-ku, Tokyo
  - CliniPro Co.,Ltd. | Tokyo-Eki Center-building Clinic - Tokyo, Japan, Chuo-ku, Tokyo
  - Minamino Cardiovascular Hospital, Hachiōji, Tokyo
  - Tokyo Angel Hospital | Clinical Trial Department, Hachiōji, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Machida Municipal Hospital, Machida, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - Tokyo Saiseikai Central Hospital | Clinical Research Center, Minato-ku, Tokyo
  - Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo
  - NewHeart Watanabe Institute, Suginami-ku, Tokyo
  - National Hospital Organization Disaster Medical Center, Tachikawa, Tokyo
  - JCHO Tokuyama Central Hospital, Shūnan, Yamaguchi
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Fukui General Clinic, Fukui
  - Fukui Prefectural Hospital, Fukui
  - Social Medical Corporation the Chiyukai foundation Fukuoka Wajiro Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Fukuoka University Nishijin Hospital, Fukuoka
  - Kyushu Central Hospital, Fukuoka
  - Gifu Heart Center, Gifu
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Tenyoukai Central Clinic, Kagoshima
  - Kagoshima Medical Center, Kagoshima
  - Chikamori Hospital, Kochi
  - Kumamoto Kinoh Hospital, Kumamoto
  - Rakuwakai Otowa Hospital, Kyoto
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Miyazaki Medical Association Hospital, Miyazaki
  - The Sakakibara Heart Institute of Okayama, Okayama
  - CMIC HealthCare Institute Co. Ltd. | Local IAA OCGMC - Okayama City Civic Hospital - Clinical Trial Centre, Okayama
  - CMIC HealthCare Institute Co. Ltd. | Okayama Rosai Hospital - Clinical Trial Centre, Okayama
  - Osaka Saiseikai Nakatsu Hospital, Osaka
  - Kitada Clinic, Osaka
  - Osaka Police Hospital | Clinical Research and Trial Center, Osaka
  - Nippon Life Hospital, Osaka
  - Japan Community Health Care Organization Osaka Hospital, Osaka
  - Oita Prefectural Hospital, Ōita
  - Saga Memorial Hospital, Saga
  - Sainokuni Higashiomiya Medical Center, Saitama
  - Sanai hospital, Saitama
  - Iwatsuki-minami Hospital, Saitama
  - Shizuoka City Shizuoka Hospital, Shizuoka
  - Saiseikai Wakayama Hospital | Pharmaceutical department, Wakayama
- Latvia (14):
  - Doctor's Practice in Cardiology, Daugavpils
  - SIA ARI Med, Daugavpils
  - Daugavpils Regional Hospital, Daugavpils
  - Rutas Eglites GP Practice, Kuldīga
  - Liepaja Regional Hospital, Liepāja
  - Lija Mora physician practice, Ogre
  - 1st Riga Clinical Hospital, Riga
  - P. Stradins Clinical University Hospital, Riga
  - Health Center Adoria, Riga
  - Health Center 4, Riga
  - Riga East Clinical University Hospital "Gailezers", Riga
  - APS Clinic, Riga
  - Vidzemes Hospital, Valmiera
  - Gita Rancane - cardiology private practice, Ventspils
- Lithuania (14):
  - Mariu klinika JSC, Kaunas
  - LUHS Kauno Hospital (Laisves ave.), Kaunas
  - LUHS Kauno Hospital (Josvainiu str.), Kaunas
  - Kardiolitos klinikos / BMP, Kaunas
  - Saules family medicine center, Kaunas
  - Hospital of LT University of Health Sciences Kaunas Clinics, Kaunas
  - InMedica clinic Zaliakalnis, Kaunas
  - Kardiologijos ir reabilitacijos klinika, Klaipėda
  - Klaipeda Republican Hospital, Klaipėda
  - Klaipeda Seamen's Hospital Cardiology Department I, Klaipėda
  - Klaipedos Jurininku Ligonine, Klaipėda
  - Siauliai Republican hospital, Šiauliai
  - InMedica Clinic Santariskes, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Malaysia (15):
  - Hospital Sultanah Bahiyah, Alor Star
  - University Hospital Kebangsaan Malaysia, Cheras
  - Hospital Sultanah Aminah, Johor Bahru
  - Hospital Raja Perempuan Zainab II, Kelantan
  - Hospital Universiti Sains Malaysia, Kelantan
  - Institute Jantung Negara, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuala Pahang
  - Hospital Al-Sultan Abdullah (UiTM Hospital), Kuala Selangor
  - Hospital Serdang, Kuala Selangor
  - Hospital Sultan Abdul Aziz Shah, Kuala Selangor
  - Hospital Seberang Jaya, Pulau Pinang
  - Sarawak General Hospital, Sarawak
  - Sarawak Heart Centre, Sarawak
  - Seremban Hospital Neurology, Seremban
- Netherlands (24):
  - Admiraal de Ruyterziekenhuis, Goes, Zeeland
  - Ziekenhuis Amstelland, Amstelveen
  - Amsterdam UMC | Heart Centre - Curius Research Department, Amsterdam
  - Gelre Apeldoorn Ziekenhuizen | Cardiology Department, Apeldoorn
  - Rijnstate | Arnhem - Cardiology Department - Cardio Research, Arnhem
  - Rode Kruis Ziekenhuis, Beverwijk
  - Tergooiziekenhuizen-Blaricum, Blaricum
  - Amphia Breda | Department of Cardiology, BMC Research, Breda
  - The Van Weel-Bethesda Hospital | Research Department, Dirksland
  - Albert Schweitzer Ziekenhuis | Dordwijk - Cardiology Department, Dordrecht
  - Catharina Hospital | Cardiology Department, Eindhoven
  - Treant locatie Scheper, Emmen
  - Medisch Spectrum Twente | Thorax Centrum Twente - Foundation Cardiovascular Research and Education Enschede, Enschede
  - Rivas | Beatrix Hospital Gorinchem - Cardiology Department, Gorinchem
  - Universitair Medisch Centrum Groningen, Groningen
  - Martini Ziekenhuis, Locatie van Swieten, Groningen
  - Spaarne Gasthuis | Haarlem Zuid - Cardiology, Haarlem
  - Saxenburgh Medisch Centrum | Cardiology Department, Hardenberg
  - Bravis Ziekenhuis | Roosendaal - Cardiology Department, Roosendaal
  - Medisch Centrum Haaglanden, Locatie Westeinde, The Hague
  - HagaZiekenhuis | Cardiology Department, The Hague
  - Ziekenhuis Rivierenland | Cardiology Research Department, Tiel
  - VieCuri - Medisch Centrum voor Noord-Limburg locatie Venlo, Venlo
  - Zaans Medisch Centrum | Hartvaatcentrum, Zaandam
- Norway (17):
  - Ålesund Sykehus, Kardiologisk Seksjon, Ålesund
  - Nordlandssykehuset Bodø Cardio, Bodø
  - Vestre Viken HF - Drammen Sykehus Cardiology, Drammen
  - Sykehuset Innlandet HF Elverum, Elverum
  - Sykehus Østfold Kalnes Cardio, Fredrikstad
  - Vestre Viken HF - Bærum Sykehus Cardiology, Gjettum
  - Sykehuset i Gjøvik Medisinsk, Gjøvik
  - UNN Harstad Medisinsk avdeling, Harstad
  - Sykehuset Lillehammer Medicine, Lillehammer
  - Molde Sjukehus Medisinsk, Molde
  - Akershus University Hospital Cardiology Department, Nordbyhagen
  - Rikshospitalet Cardiology, Oslo
  - Diakonhjemmets sykehus, Oslo
  - OUS Ullevål Cardiology, Oslo
  - Skedsmo Medisinske Senter, Skedsmokorset
  - Stavanger UHospital Cardiology, Stavanger
  - UNN Tromsø Cardiology Dep., Tromsø
- Poland (26):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - KLIMED Marek Klimkiewicz, Bialystok
  - MICS Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Centrum Medyczne KerMed, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Samodzielny Publiczny Specjalistyczny Szpital Zachodni, Grodzisk Mazowiecki
  - CLINICAL MEDICAL RESEARCH Sp. z o. o., Katowice
  - Vita Longa Sp. z o.o., Katowice
  - Unicardia Specjalistyczne Centrum Leczenia Ch.Serca i Naczyn, Krakow
  - Centrum Terapii Wspolczesnej, Lodz
  - CM MED-GASTR Sp. z o.o., Lodz
  - Centrum Medyczne Ogrodowa G. i M. Kania Lekarze i Lekarze Dentysci Spólka Partnerska z siedziba w Skierniewicach, Lowicz
  - 1 Wojskowy Szpital Kliniczny z Poliklinika SPZOZ w Lublinie, Lublin
  - NZOZ "Twoja Przychodnia" Sp. z o.o., Lublin
  - Futuremeds sp. z o. o., Olsztyn
  - Etyka Osrodek Badan Klinicznych, Olsztyn
  - NZOZ Heureka, Piaseczno
  - Irmed Klimkiewicz, Rudziewicz-Kowalska Sp.j., Piotrkow Trybunalski
  - Solumed Centrum Medyczne, Poznan
  - Velocity Pulawy, Puławy
  - EMED Centrum Uslug Medycznych, Rzeszów
  - ClinMedica Research Sp. z o.o., Skierniewice
  - "Nowe Zdrowie-Ck" Kieltucki I Wspolnicy Spolka Jawna, Staszów
  - NBR Polska Tomasz Klodawski, Warsaw
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji, Warsaw
  - KO-MED Centra Kliniczne Zamosc, Zamość
- Portugal (18):
  - Hospital da Senhora da Oliveira | Clinical Research Department, Guimaraes, Braga, Braga District
  - Centro Hospitalar Universitario Cova de Beira | Clinical Research Department, Covilha, Castelo Branco District
  - Luz Saude | Hospital da Luz Lisboa - Centro de Investigacao Clinica, Lisbon, Lisbon District
  - Centro Hospitalar Universitario de Lisboa Norte | Heart and Vessels Department, Lisbon, Lisbon District
  - Hospital de Vila Franca de Xira | Centro de Desenvolvimento e Investigacao, Vila Franca de Xira, Lisbon District
  - Hospital Pedro Hispano | Clinical Research Center, Matosinhos Municipality, Porto District
  - Ucardio | Cardiology Department, Riachos, Santarém District
  - Hospital Garcia de Orta | Research Department, Almada, Setúbal District
  - Centro Clinico Academico Braga | Braga, Portugal, Braga
  - Centro Hospitalar e Universitario de Coimbra, E.P.E. | Department of Cardiology, Research Unit, Coimbra
  - Centro Hospitalar de Tamega e Sousa | Hospital Padre Americo - Cardiology Department, Guilhufe
  - Centro Hospitalar de Leiria | Santo Andre Hospital - Research Center, Leiria
  - Centro Hospitalar de Lisboa Ocidental | Clinical Research Department, Lisbon
  - Lusiadas | Hospital Lusiadas Lisboa - Lusiadas Knowledge Center, Lisbon
  - Centro Hospitalar Universitario de Sao Joao | Polo Porto - Centro de Investigacao e Ensaios Clinicos, Porto
  - Centro Hospitalar Vila Nova de Gaia e Espinho | Unit 1 - Clinical Research Center, Porto
  - Luz Saude | Hospital da Luz Setubal - Clinical Research Department, Setúbal
  - Centro Hospitalar De Tras os Montes e Alto Douro | Hospital Sao Pedro - Centro de Investigacao Clinica, Vila Real
- Romania (21):
  - Cardiomed S.R.L, Cluj-Napoca, Dolj
  - CMI. Dr. Podoleanu Cristian, Târgu Mureş, Mureș County
  - Municipal Clinical Emergency Hospital of Timisoara, Timișoara, Timiș County
  - Sp. Judetean de Urgenta Dr. Constantin Opris Baia Mare, Baia Mare
  - S.C Thera Card S.R.L, Brasov
  - S.C. Centrul Medical de Diagnostic si Tratament Ambulator Neomed SRL, Brasov
  - Emergency County Hospital, Braila, Brăila
  - Spitalul Clinic Colentina, Bucharest
  - Emergency Institute for Cardiovascular Diseases, Bucharest
  - Spitalul Clinic de Urgenta Sf. Ioan, Bucharest
  - Spitatul Universitar de Urgenta Bucaresti, Bucharest
  - Niculae Stancioiu Heart Institute Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic de Recuperare Cluj-Napoca, Cluj-Napoca
  - Sfantul Spiridon Emergency Clinical County Hospital, Iași
  - S.C. CARDIOMED S.R.L. Iasi, Iași
  - S.C. Sal Med SRL, Piteşti
  - Spitalul Judetean de Urgenta Satu Mare, Satu Mare
  - Spitalul de urgenta Sf. Ioan Cel Nou, Suceava
  - S.C. Cardio Med S.R.L., Târgu Mureş
  - Emergency Institute of Cardiovascular Diseases & Transplant, Târgu Mureş
  - Timisoara Institute of Cardiovascular Diseases, Timișoara
- Singapore (7):
  - National University Hospital, Singapore
  - National Heart Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
  - SingHealth Polyclinics - Pasir Ris, Singapore
  - Changi General Hospital, Singapore
  - Sengkang General Hospital, Singapore
  - Ng Teng Fong General Hospital, Singapore
- Slovakia (21):
  - ALIAN s.r.o., Bardejov
  - GALENUM s.r.o., Bratislava
  - Kardiosanus | Bratislava, Slovakia, Bratislava
  - Nemocnica s poliklinikou Brezno, n.o., Brezno
  - KARDIO R s.r.o., Košice
  - Medical Group Kosice s.r.o. | Kosice, Slovakia, Košice
  - KARDIO-ANGIO s.r.o., Levice
  - KardioLEV s.r.o., Levoča
  - Internal and Diabetes Clinic - IN-DIA s.r.o. | Lucenec, Slovakia, Lučenec
  - KardioMed | Outpatient Cardiology and Internal Medicine II Clinic, Lučenec
  - KARDIO 1 | Lucenec, Slovakia, Lučenec
  - ORALEK, s.r.o., Námestovo
  - Kardiocentrum Nitra | Cardiology Clinic - Outpatient Department, Nitra
  - Specializovana nemocnica sv. Svorada Zobor, n.o., Nitra
  - KaCH, s.r.o., Nové Zámky
  - BENIMED s.r.o., Piešťany
  - Medikard | Department of Internal Medicine, Prešov
  - MEDISPOL s.r.o., Prešov
  - Interna SK s.r.o., Svidník
  - Kardiologicka ambulancia Trnava, MUDr. Vladimir Macek, Trnava
  - Medivasa s.r.o., Žilina
- South Korea (20):
  - Pusan National University Hospital, Busan, Busan Gwang''yeogsi
  - Kyungpook National University Hospital, Daegu, Daegu Gwang''yeogsi
  - Yonsei University Wonju Christian Hospital, Wŏnju, Gang''weondo
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggido
  - Bundang Cha Hospital, Seongnam-si, Gyeonggido
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul, Gyeonggido
  - Ajou University Hospital, Suwon, Gyeonggido
  - Uijeongbu ST. Mary's Hospital, Uijeongbu-si, Gyeonggi-do, Gyeonggido
  - The Catholic Univ. of Korea Eunpyeong St. Mary's Hospital, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Dong-A University Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (23):
  - Complejo Hospitalario Universitario de Ferrol | Hospital Naval - Unidad de Hipertensión Arterial, Ferrol, A Coruña
  - Hospital Clinico Universitario de Santiago de Compostela | Cardiology Department, Santiago de Compostela, A Coruña
  - Hospital Universitari de Bellvitge | Bellvitge Biomedical Research Institute - Cardiology - AF, Stroke Prevention, L'Hospitalet de Llobregat, Barcelona
  - Jose Manuel Pascual Pascual S.A. | Hospital Virgen del Camino - Internal Medicine Department, Sanlúcar de Barrameda, Cádiz
  - Jose Manuel Pascual Pascual S.A. | Hospital Virgen de las Montanas - Internal Medicine Department, Villamartín, Cádiz
  - Hospital Universitario de La Princesa | Internal Medicine Department, Madrid, Madrid [es-m]
  - Hospital Universitario Virgen de la Victoria | Cardiology Department, Málaga, Málaga
  - Hospital Universitario Central de Asturias | Servicio de Cardiologia, Oviedo, Principality of Asturias
  - Hospital Alta Resolucion de Lebrija | Cardiology Service Department, Lebrija, Sevilla
  - Hospital Alta Resolucion de Utrera | Cardiology Service Department, Utrera, Sevilla
  - University Hospital of A Coruna | Cardiology department, A Coruña
  - Hospital General Universitario Doctor Balmis de Alicante | Cardiology Department, Alicante
  - Hospital de la Santa Creu i Sant Pau | Cardiology Department, Barcelona
  - Vall d'Hebron Barcelona Hospital Campus | Vall d'Hebron Hospital Universitario - Cardiology Department, Barcelona
  - Hospital Quironsalud Barcelona | Internal Medicine Department, Barcelona
  - Hospital Universitario Ramon y Cajal | Departamento de Medicina Interna, Madrid
  - Hospital Universitario 12 de Octubre | Cardiology Department, Madrid
  - Hospital Universitario La Paz | Cardiology Department - AF, Stroke Prevention, Madrid
  - Hospital Universitario La Paz | IdiPAZ - Neurology Department, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca | Cardiology Department, Murcia
  - Hospital Universitario Virgen del Rocio | Hospital General - Departamento de Cardiologia y Cirugia Cardiovascular, Seville
  - Hospital General Universitario de Valencia | Cardiology Department, Valencia
  - La Fe University and Polytechnic Hospital | Cardiology Department, Valencia
- Sweden (18):
  - Södra Älvsborgs Sjukhus, Borås
  - Falu Lasarett, Falun
  - SU/Östra, Gothenburg
  - Helsingborgs Lasarett, Helsingborg
  - Universitetssjukhuset i Linköping, Linköping
  - Clemenstorget Hjärtmottagning, Lund
  - Skånes Universitetssjukhus, Lund
  - SU/Mölndal, Mölndal
  - Vrinnevisjukhuset, Norrköping
  - Universitetssjukhuset Örebro, Örebro
  - Skellefteå Lasarett, Skellefteå
  - Södersjukhuset AB, Stockholm
  - Karolinska Universitetssjukhuset Huddinge Stockholm, Stockholm
  - Karolinska Universitetssjukhuset, Stockholm
  - Danderyds sjukhus, Stockholm
  - Norrlands Universitetssjukhus, Umea, Umeå
  - Akademiska Sjukhuset, Uppsala
  - Västmanlands Sjukhus Västerås, Västerås
- Switzerland (7):
  - Kantonsspital Aarau, Aarau, Canton of Aargau
  - Kantonsspital Baden, Baden, Canton of Aargau
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Inselspital Universitätsspital Bern, Bern
  - Cardiocentro Ticino, Lugano
  - UniversitätsSpital Zürich, Zurich
- Taiwan (23):
  - National Yang Ming Chiao Tung University Hospital, Yilan, Ilan
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung
  - Chi Mei Medical Center, Taikang, Tainan
  - MacKay Memorial Hospital Tamsui Branch, New Taipei City, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei, Taipei
  - Changhua Christian Hospital, Changhua
  - Mackay Memorial Hospital - Hsinchu Branch, Hsinchu
  - Buddhist Tzu-Chi General Hospital, Hualien, Hualien City
  - Veterans General Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Medical University | Clinical Research Center, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District
- Turkey (Türkiye) (17):
  - Afyonkarahisar Saglik Bilimleri Universitesi, Afyonkarahisar
  - Baskent Universitesi Tip Fakultesi Hastanesi, Ankara
  - Health Ministry Of Türkiye Republic Ankara Bilkent City Hospital, Ankara
  - Akdeniz Universitesi Tip Fakultesi Hastanesi, Antalya
  - Hitit Universitesi Tip Fakultesi, Çorum
  - Ataturk Universitesi Tip Fakultesi, Erzurum
  - Eskisehir Osmangazi Universitesi Tip Fakultesi, Eskişehir
  - Istanbul Universitesi Cerrahpasa - Kardiyoloji Anabilim Dali, Istanbul
  - Marmara Uni. Tip Fak. Pendik EAH Kardiyoloji, Istanbul
  - Istanbul Mehmet Akif Ersoy Gogus Kalp Damar Cerrahisi E.A.H., Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
  - Izmir Ekonomi Universitesi Medikal Point Hastanesi, Izmir
  - Erciyes Universitesi Tip Fakultesi, Kayseri
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Kutahya Saglik Bilimleri Uni. Evliya Celebi Egitim ve Arasti, Kütahya
  - Adana Sehir Egitim ve Arastirma Hastanesi, Medreseboğazı
  - Saglik Bilimleri Univ. Samsun EAH Kardiyoloji Departmani, Samsun
- United Kingdom (24):
  - Staploe Medical Centre, Ely, Cambridgeshire
  - Countess of Chester Hospital, Chester, Cheshire
  - Chesterfield Royal Hospital, Chesterfield, Derbyshire
  - Torbay Hospital, Torbay, Devon
  - Poole Hospital NHS Trust, Poole, Dorset
  - Glasgow Royal Infirmary | Stroke Unit, Glasgow, Glasgow City
  - North Hampshire Hospital, Basingstoke, Hampshire
  - Lister Hospital, Stevenage, Hertfordshire
  - Queen Elizabeth the Queen Mother Hospital, Margate, Kent
  - University Hospitals Leicester, Leicester, Leicestershire
  - Northwick Park Hospital, Harrow, London
  - Charing Cross Hospital, London, London
  - Craigavon Area Hospital, Craigavon, North Ireland
  - Wansbeck General Hospital, Ashington, Northumberland
  - Freeman Hospital, Newcastle, Tyne and Wear
  - Soho Health Centre, Future Meds, Birmingham, West Midlands
  - Russells Hall Hospital, Dudley, West Midlands
  - St Richard's Hospital, Chichester, West Sussex
  - Worcestershire Acute Hospital Trust, Worcester, Worcestershire
  - James Cook University Hospital South Tees, Middlesbrough, Yorkshire
  - Ely Bridge Medical Centre, Cardiff
  - Heart and Chest Hospital, Liverpool
  - King's College Hospital - NHS Foundation Trust, London
  - Future Meds - Bromborough, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Alexander JH, Lydon EJ, Piccini JP, Viethen T, Oldgren J, Goodman SG, Steffel J, Russo AM, van Gelder IC, Ferdinand KC, Lopes RD, Mundl H, Benczur B, Gomez-Doblas JJ, Glikson M, Goudev A, Grove EL, Halvorsen S, Kiviniemi T, Martin AC, Sandhu RK, Vinereanu D, Rockhold FW, Caso V, Coppolecchia R, Patel MR. Asundexian or Apixaban in Patients With Atrial Fibrillation According to Prior Oral Anticoagulant Use: A Subgroup Analysis of the OCEANIC-AF Randomized Clinical Trial. JAMA Cardiol. 2025 Jun 1;10(6):555-563. doi: 10.1001/jamacardio.2025.0277. PMID 40136309
- [Derived] Piccini JP, Patel MR, Steffel J, Ferdinand K, Van Gelder IC, Russo AM, Ma CS, Goodman SG, Oldgren J, Hammett C, Lopes RD, Akao M, De Caterina R, Kirchhof P, Gorog DA, Hemels M, Rienstra M, Jones WS, Harrington J, Lip GYH, Ellis SJ, Rockhold FW, Neumann C, Alexander JH, Viethen T, Hung J, Coppolecchia R, Mundl H, Caso V; OCEANIC-AF Steering Committee and Investigators. Asundexian versus Apixaban in Patients with Atrial Fibrillation. N Engl J Med. 2025 Jan 2;392(1):23-32. doi: 10.1056/NEJMoa2407105. Epub 2024 Sep 1. PMID 39225267
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/19767

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 1035 study centers across in Asia, Europe, North America, South America, and Australia, between 05-Dec-2022 (first participant first visit) and 31-Jan-2024 (last participant last visit).
Pre-assignment Details: A total of 16436 participants were screened, of whom 1606 participants were screen failures. 14830 of the screened participants were randomized to treatment and 14757 participants were treated. 73 participants never received study intervention.
Groups:
- Asundexian: Participants received asundexian 50 mg once a day (OD) and apixaban matching placebo.
- Apixaban: Participants received apixaban 5 mg twice a day (BID) or reduced dose 2.5 mg BID and asundexian matching placebo.
Period: Overall Study
Arm/Group | Asundexian | Apixaban
Started | 7383 | 7374
Completed | 6901 | 7012
Not Completed | 482 | 362
Not completed — Adverse Event | 117 | 90
Not completed — Death | 53 | 57
Not completed — Lost to Follow-up | 6 | 3
Not completed — Other | 18 | 15
Not completed — Outcome event | 64 | 36
Not completed — Physician Decision | 33 | 19
Not completed — Protocol-specified withdrawal criterion met | 2 | 2
Not completed — Site terminated by sponsor | 10 | 10
Not completed — Study terminated by sponsor | 1 | 0
Not completed — Withdrawal by Subject | 178 | 130

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All participants randomized to study intervention including participants who did not receive study intervention. N (number) =14830 Adjusted Full Analysis Set (aFAS): All participants in the Full Analysis Set excluding subjects randomized from one site in Japan. N=14810 Due to Good Clinical Practice violations, 20 participants from one site in Japan were excluded from all analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Asundexian | Apixaban | Total
Number analyzed (Participants) | 7415 | 7395 | 14810
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.9 (7.7) | 73.9 (7.7) | 73.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2656 | 2558 | 5214
  Male | 4759 | 4837 | 9596
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 533 | 507 | 1040
  Not Hispanic or Latino | 6774 | 6793 | 13567
  Unknown or Not Reported | 108 | 95 | 203
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 2035 | 2010 | 4045
  Native Hawaiian or Other Pacific Islander | 9 | 2 | 11
  Black or African American | 88 | 95 | 183
  White | 5216 | 5211 | 10427
  More than one race | 21 | 28 | 49
  Unknown or Not Reported | 42 | 45 | 87

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite of Stroke or Systemic Embolism
Description: The assessment was based on the cause-specific hazard ratio (csHR), comparing asundexian with apixaban which is based on time to first event.
  Stroke was defined as an acute episode of focal or global neurological dysfunction caused by an injury of the brain, spinal cord, or retina as a result of hemorrhage or infarction.
  Systemic embolism is defined as abrupt vascular insufficiency associated with clinical or radiological evidence of arterial occlusion in the absence of other likely mechanisms (this does not include myocardial infarction, thromboembolism of the pulmonary vasculature or venous thrombosis, e.g. pulmonary embolism or deep venous thrombosis).
Time Frame: Approximately 12 months
Population: aFAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7415 | 7395
Participants | 98 | 26
Statistical Analysis 1: Comparison: Asundexian vs Apixaban; Comparison of Asundexian 50 mg verus Apixaban; Test type: Superiority; p < .0001, Log Rank; Cox Proportional Hazard = 3.785, 95% CI 2-sided [2.457 to 5.833]
Statistical Analysis 2: Comparison: Asundexian vs Apixaban; Comparison of Asundexian 50 mg verus Apixaban; Test type: Superiority; p < .0001, Gray's test; Fine-Gray model = 3.790, 95% CI 2-sided [2.460 to 5.839]

2. Primary Outcome: Number of Participants With International Society on Thrombosis and Hemostasis (ISTH) Major Bleeding
Description: Assessment based on the (csHR), comparing asundexian with apixaban which is based on time to first event.
  ISTH Major Bleeding was defined as an event that meets at least one of the below criteria, based on the definition given by the ISTH (Schulman and Kearon 2005):
  * Fatal bleeding, and/or
  * Symptomatic bleeding in a critical area or organ (intracranial, intraspinal, intraocular with compromised vision, pericardial, retroperitoneal, intra-articular, or intramuscular with compartment syndrome), and/or
  * Clinically overt* bleeding associated with a recent (within 48 hours) decrease in the hemoglobin level of ≥ 2 g/dL (20 g/L; 1.24 mmol/L) compared with the most recent hemoglobin value available before the event, and/or
  * Clinically overt* bleeding leading to transfusion of 2 or more units of packed red blood cells or whole blood.
    * Overt bleeding required the identification of the bleeding location and the hemoglobin drop and/or transfusion needed to be related to the bleeding.
Time Frame: Approximately 12 months
Population: Safety Analysis Set (SAF): All participants randomized to study intervention and who took at least 1 dose of study intervention. N=14757 Adjusted Safety Analysis Set (aSAF): All participants in the Safety Analysis Set excluding subjects randomized from one site in Japan. N=14737 Due to Good Clinical Practice violations, 20 participants from one site in Japan were excluded from all analyses.
  aSAF population was analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7373 | 7364
Participants | 17 | 53
Statistical Analysis 1: Comparison: Asundexian vs Apixaban; Comparison of Asundexian 50 mg verus Apixaban; Test type: Superiority; p < .0001, Log Rank; Fine-Gray model = 0.319, 95% CI 2-sided [0.185 to 0.552]
Statistical Analysis 2: Comparison: Asundexian vs Apixaban; Comparison of Asundexian 50 mg verus Apixaban; Test type: Superiority; p < .0001, Gray's test; Fine-Gray model = 0.316, 95% CI 2-sided [0.182 to 0.547]

3. Primary Outcome: Number of Participants With Composite of Stroke, Systemic Embolism, or ISTH Major Bleeding
Description: The assessment was based on the cause-specific hazard ratio (csHR), comparing asundexian with apixaban which is based on time to first event.
Time Frame: Approximately 12 months
Population: aSAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7373 | 7364
Participants | 120 | 75
Statistical Analysis 1: Comparison: Asundexian vs Apixaban; Comparison of Asundexian 50 mg verus Apixaban; Test type: Superiority; p = 0.0011, Log Rank; Fine-Gray model = 1.610, 95% CI 2-sided [1.207 to 2.149]
Statistical Analysis 2: Comparison: Asundexian vs Apixaban; Comparison of Asundexian 50 mg verus Apixaban; Test type: Superiority; p = 0.0013, Gray's test; Fine-Gray model = 1.599, 95% CI 2-sided [1.197 to 2.134]

4. Secondary Outcome: Number of Participants With Composite of Ischemic Stroke or Systemic Embolism
Description: The assessment was based on the cause-specific hazard ratio (csHR), comparing asundexian with apixaban which is based on time to first event.
  An ischemic stroke was defined as the rapid onset (or present on awakening) of a new focal neurological deficit with clinical (> 24 hours symptoms / signs) or imaging evidence of infarction that is not attributable to a non-ischemic cause (i.e. not associated with infection, tumor, seizure, severe metabolic disease).
Time Frame: Approximately 12 months
Population: aFAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7415 | 7395
Participants | 96 | 22

5. Secondary Outcome: Number of Participants With All-cause Mortality
Description: as for outcome 3
Time Frame: Approximately 12 months
Population: aFAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7415 | 7395
Participants | 60 | 71

6. Secondary Outcome: Number of Participants With Ischemic Stroke
Description: as for outcome 4
Time Frame: Approximately 12 months
Population: aFAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7415 | 7395
Participants | 85 | 21

7. Secondary Outcome: Number of Participants With Cardiovascular (CV) Death
Description: The assessment was based on the cause-specific hazard ratio (csHR), comparing asundexian with apixaban which is based on time to first event.
  CV death included death due to stroke, myocardial infarction, heart failure or cardiogenic shock, sudden death or any other death due to other cardiovascular causes or CV procedures. In addition, death due to non-traumatic cardiovascular hemorrhage will be included, e.g. non-stroke intracranial hemorrhage, non-procedural or non-traumatic vascular rupture (e.g. aortic aneurysm), or hemorrhage causing cardiac tamponade
Time Frame: Approximately 12 months
Population: aFAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7415 | 7395
Participants | 48 | 44

8. Secondary Outcome: Number of Participants With Composite of CV Death, Stroke, or Myocardial Infarction (MI)
Description: The assessment was based on the cause-specific hazard ratio (csHR), comparing asundexian with apixaban which is based on time to first event.
  The diagnosis of MI requires the combination of:
  * Presence of acute myocardial injury (changes in cardiac biomarkers) and
  * Evidence of acute myocardial ischemia derived from the clinical presentation, electrocardiographic changes, or the results of myocardial or coronary artery imaging, or in case of post mortem pathological findings irrespective of biomarker values.
Time Frame: Approximately 12 months
Population: aFAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7415 | 7395
Participants | 155 | 77

9. Secondary Outcome: Number of Participants With Composite of ISTH Major or Clinically Relevant Non-major Bleeding
Description: The assessment was based on the cause-specific hazard ratio (csHR), comparing asundexian with apixaban which is based on time to first event.
  Clinically relevant non-major bleeding was considered any sign or symptom of acute or sub-acute clinically overt bleeding that does not fit the criteria for the ISTH definition of major bleeding, but does meet at least one of the following criteria (based on criteria published by the EMA) (EMA 2014):
  * requiring medical or surgical treatment by a healthcare professional for bleeding
  * leading to hospitalization or increased level of care for bleeding
  * a change in antithrombotic therapy (including study intervention) for bleeding *Overt bleeding required the identification of the bleeding location.
Time Frame: Approximately 12 months
Population: aSAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7373 | 7364
Participants | 83 | 188

10. Secondary Outcome: Number of Participants With Clinically Relevant Non-major Bleeding
Description: as for outcome 3
Time Frame: Approximately 12 months
Population: aSAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7373 | 7364
Participants | 67 | 140

11. Secondary Outcome: Number of Participants With Hemorrhagic Stroke
Description: The assessment was based on the cause-specific hazard ratio (csHR), comparing asundexian with apixaban which is based on time to first event.
  Hemorrhagic stroke was defined as an acute, atraumatic extravasation of blood into the brain parenchyma, intraventricular or subarachnoid space with associated neurological symptoms. This does not include microbleeds or hemorrhagic transformation of an ischemic stroke.
Time Frame: Approximately 12 months
Population: aSAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7373 | 7364
Participants | 1 | 6

12. Secondary Outcome: Number of Participants With Intracranial Hemorrhage
Description: as for outcome 3
Time Frame: Approximately 12 months
Population: aSAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7373 | 7364
Participants | 3 | 18

13. Secondary Outcome: Number of Participants With Fatal Bleeding
Description: as for outcome 3
Time Frame: Approximately 12 months
Population: aSAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7373 | 7364
Participants | 0 | 4

14. Secondary Outcome: Number of Participants With Minor Bleeding
Description: The assessment was based on the cause-specific hazard ratio (csHR), comparing asundexian with apixaban which is based on time to first event.
  All other overt bleeding episodes not meeting the criteria for ISTH major or clinically relevant non-major bleeding were classified as minor bleeding (for example, bleeding from a minor wound that does not prompt a treatment for the bleeding, for instance with surgical hemostasis, or epistaxis that does not require a medical treatment for bleeding or a change in antithrombotic therapy).
Time Frame: Approximately 12 months
Population: aSAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7373 | 7364
Participants | 187 | 317

15. Secondary Outcome: Number of Participants With Composite of Stroke, Systemic Embolism, ISTH Major Bleeding, or All-cause Mortality
Description: as for outcome 3
Time Frame: Approximately 12 months
Population: aSAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7373 | 7364
Participants | 149 | 101

16. Secondary Outcome: Number of Participants With Composite of Disabling Stroke (mRS ≥ 3), Critical Bleeding, or All-cause Mortality
Description: The assessment was based on the cause-specific hazard ratio (csHR), comparing asundexian with apixaban which is based on time to first event.
  Critical bleeding was defined as symptomatic bleeding in either of the following critical locations (intracranial, intraspinal, pericardial, intra-articular, or retroperitoneal) or as intraocular bleeding with compromised vision or intramuscular bleeding with compartment syndrome.
Time Frame: Approximately 12 months
Population: aSAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian | Apixaban
Number analyzed (Participants) | 7373 | 7364
Participants | 51 | 56

ADVERSE EVENTS:
Time Frame: Approximately 12 months
Description: AEs that occurred or worsened after the first dose of study intervention up to 2 days after the last dose of study intervention are considered treatment-emergent. Adverse event reporting for the all-cause mortality considers all deaths that occurred at any time during the study before the last contact.
Arm/Group | Asundexian | Apixaban
All-Cause Mortality (participants affected / at risk) | 73/7373 | 85/7364
Serious Adverse Events (participants affected / at risk) | 582/7373 | 599/7364
Other Adverse Events (participants affected / at risk) | 467/7373 | 455/7364
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asundexian (N=7373) | Apixaban (N=7364)
Anaemia (Blood and lymphatic system disorders) | 5 (7) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 4 (4) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 4 (4) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 47 (50) | 71 (84)
Atrial flutter (Cardiac disorders) | 8 (8) | 5 (5)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 4 (4) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 6 (7) | 8 (9)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 54 (55) | 62 (78)
Cardiac failure acute (Cardiac disorders) | 18 (23) | 25 (28)
Cardiac failure chronic (Cardiac disorders) | 18 (18) | 8 (8)
Cardiac failure congestive (Cardiac disorders) | 10 (13) | 14 (15)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 2 (2)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 6 (7) | 5 (5)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (2) | 3 (3)
Low cardiac output syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 2 (2)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 2 (2) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinoatrial block (Cardiac disorders) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (3) | 3 (3)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 6 (6) | 3 (5)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Dilated cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 2 (2)
Acute left ventricular failure (Cardiac disorders) | 3 (3) | 5 (5)
Arrhythmic storm (Cardiac disorders) | 1 (1) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 3 (3) | 5 (5)
Chronic coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (5) | 4 (4)
Vertigo labyrinthine (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Thyrotoxic crisis (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 3 (3)
Eyelid ptosis (Eye disorders) | 1 (1) | 1 (1)
Pseudopapilloedema (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Epiretinal membrane (Eye disorders) | 1 (1) | 1 (1)
Rhegmatogenous retinal detachment (Eye disorders) | 2 (2) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 6 (6)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 6 (6) | 5 (5)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Melaena (Gastrointestinal disorders) | 2 (2) | 5 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 3 (3) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 11 (11) | 11 (11)
Chills (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 6 (6) | 5 (5)
Gait disturbance (General disorders) | 3 (3) | 1 (1)
Mass (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 4 (4)
Sudden death (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 2 (2) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Gait deviation (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Medical device site haematoma (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 2 (2)
Procedural failure (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 5 (5) | 3 (3)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 0 (0) | 1 (1)
Congestive hepatopathy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1)
Cellulitis (Infections and infestations) | 9 (10) | 3 (4)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1)
Cryptosporidiosis infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 1 (1)
Cystitis escherichia (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 2 (3) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 2 (2)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4)
Meningitis listeria (Infections and infestations) | 0 (0) | 1 (1)
Nosocomial infection (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 2 (2)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 22 (22) | 28 (34)
Pneumonia aspiration (Infections and infestations) | 4 (4) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 3 (3)
Septic shock (Infections and infestations) | 2 (2) | 5 (5)
Skin infection (Infections and infestations) | 3 (3) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 7 (7) | 13 (14)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 4 (4)
Rectal abscess (Infections and infestations) | 1 (1) | 1 (1)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess soft tissue (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 (7) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Enterocolitis bacterial (Infections and infestations) | 2 (2) | 0 (0)
Chikungunya virus infection (Infections and infestations) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1)
Bullous erysipelas (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 7 (7) | 10 (10)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Klebsiella urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Femur fracture (Injury, poisoning and procedural complications) | 9 (9) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Colonoscopy (Investigations) | 1 (1) | 0 (0)
Endoscopy upper gastrointestinal tract (Investigations) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Scan myocardial perfusion abnormal (Investigations) | 1 (1) | 0 (0)
Clostridium test positive (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Hypervolaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (6)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Still's disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral lateral recess stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Meniscopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chordoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Extramammary Paget's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Appendix adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
High-grade B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bing-Neel syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral circulatory failure (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Motor neurone disease (Nervous system disorders) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2)
Sciatica (Nervous system disorders) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 3 (3)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 10 (11) | 12 (13)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic transformation stroke (Nervous system disorders) | 2 (2) | 0 (0)
Putamen haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Postresuscitation encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cervicogenic vertigo (Nervous system disorders) | 1 (2) | 0 (0)
Post stroke epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial mass (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Neuropsychological symptoms (Psychiatric disorders) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 5 (6)
Nephrolithiasis (Renal and urinary disorders) | 5 (5) | 2 (2)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 2 (2)
Urinary retention (Renal and urinary disorders) | 4 (4) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 1 (1)
Nephritic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 26 (26) | 12 (12)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (7)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 11 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough variant asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abstains from alcohol (Social circumstances) | 0 (0) | 1 (2)
Aortic stenosis (Vascular disorders) | 3 (3) | 3 (3)
Haematoma (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 5 (6)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 3 (3)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (2) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (3) | 1 (1)
Hypoperfusion (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1)
Aortic rupture (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 3 (3)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Vein dissection (Vascular disorders) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asundexian (N=7373) | Apixaban (N=7364)
Diarrhoea (Gastrointestinal disorders) | 115 (124) | 72 (73)
Nasopharyngitis (Infections and infestations) | 98 (104) | 89 (92)
COVID-19 (Infections and infestations) | 97 (99) | 109 (109)
Dizziness (Nervous system disorders) | 132 (138) | 113 (120)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 50 (59) | 96 (120)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT05643573/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT05643573/SAP_001.pdf